CLINICAL TRIAL: NCT00780975
Title: A Phase II, Multicenter, Open-label, Clinical and Pharmacokinetic Study of Aplidin® as a 3-hour IV Infusion Every 2 Weeks, in Relapsing or Refractory Patients With Androgen-independent Prostate Adenocarcinoma..
Brief Title: A Study of Aplidin ( Plitidepsin) in Subjects With Advanced Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-B-011-02
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: Aplidin; Plitidepsin; Prostate; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — plitidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Aplidin (Plitidepsin)
  Interventions: Drug: Aplidin (plitidepsin)

INTERVENTIONS:
Drug: Aplidin (plitidepsin) — Aplidin® administered at a starting dose of 5 mg/m2, as a 3-hours intravenous infusion, every 2 weeks.

SUMMARY:
This is a study to test the safety and efficacy of an investigational chemotherapy agent in patients with advanced prostate cancer. Subjects who meet all entry criteria and have signed the informed consent will be enrolled in the study. Participants will be required to attend regular clinic visits to receive study medication and have their status monitored. A detailed explanation can be provided by the investigator conducting the study.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-cutaneous cancer diagnosed in men in the United States. The majority of deaths occur in men with androgen-independent prostate cancer [AIPC]. Although 80% of men with advanced cancer will initially respond to androgen ablation with disease regression or stabilization, their malignancies become resistant to such therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before starting any study-specific procedure. If any patient is unable to give consent, it may be obtained from the patient's legal representative if in accordance with local laws and regulations.
2. Men with castrate metastatic adenocarcinoma of the prostate, with the following characteristics:

   * Confirmed pathological diagnosis.
   * Metastatic disease (radiologically documented).
   * All patients with chemical castration must have a serum testosterone level below 50 ng/ml. There is no need to document a serum testosterone in patients having a prior surgical castration2.
   * Baseline PSA > 5 ng/ml (according to the recommendations from the Prostate-Specific Antigen Working Group2).
   * Androgen-independent progressive disease, as defined by detectable, rising PSA in two consecutive measurements at least one week apart:

     * If PSA responded to a prior therapy, progression occurs when the PSA is 50% above the nadir level.
     * If PSA did not respond to a prior therapy, progression occurs when the PSA increases by 25% or more above pretreatment levels.
     * In both cases, the increase in absolute value PSA level must be at least 5 ng/ml, and must be confirmed by a second measurement a minimum of 1 week later.
   * Patients must have received prior docetaxel-based chemotherapy.
3. Recovery from any toxicity derived from previous treatments. The presence of alopecia and NCI-CTC grade < 2 sensitive peripheral neuropathy is allowed.
4. Age > 18 years.
5. Performance status (ECOG) < 2.
6. Life expectancy > 3 months.
7. Adequate renal, hepatic, and bone marrow function (assessed < 14 days before inclusion in the study):

   * Neutrophil count ³ 1.5 x 109/L.
   * Platelet count ³ 100 x 109/L. Hemoglobin > 9 g/dl.
   * Creatinine clearance ³ 40 ml/min (calculated from the Cockcroft and Gault formula), see Appendix 3.
   * Serum bilirubin * 1.5 mg/dl.
   * AST, ALT < 2.5 x ULN (< 5 x ULN in case of liver metastasis).
   * Albumin > 25 g/L.
8. Left ventricular ejection fraction within normal limits

Exclusion Criteria:

1. Prior therapy with Aplidin®.
2. Concomitant therapy with any anti-tumor agent, including glucocorticoids at a daily dose greater than 10 mg prednisone or equivalent, except when they were indicated for symptom control, provided that disease progression was documented while on steroids.
3. Small cell carcinoma of the prostate.
4. More than two previous lines of systemic therapy for patient's castrate metastatic disease, considering biological agents or chemotherapy as systemic therapy.
5. Patients with progressive measurable disease but without increased PSA value (according to the consensus recommendations) will not be considered eligible.
6. Wash-out periods less than:

   * 6 weeks after the last dose of a nitroso-urea or high dose chemotherapy
   * 4 weeks after the last dose of other chemotherapies or biological agents
   * 6 weeks after the end of treatment with extensive external beam radiation (more than 25% of bone marrow distribution) or radionuclide therapy.
   * 4 weeks after the end of treatment with palliative radiation involving less than 25% of bone marrow reserves.
   * 4 weeks for major prior surgery
   * 30 days after receiving any other investigational product
7. Men of reproductive potential who are not using effective contraceptive methods, considering complete abstinence from intercourse throughout the treatment with the study drug and for at least 6 months after completion or premature discontinuation from the study as an effective contraceptive method, to be sure that the patient's female partner does not become pregnant.
8. History of another neoplastic disease. The exceptions are:

   8.1 Non-melanoma skin cancer. 8.2 Any other cancer curatively treated with no evidence of disease for at least 10 years.
9. Known symptomatic cerebral or leptomeningeal involvement.
10. Other relevant diseases or adverse clinical conditions:

    * History or presence of unstable angina, myocardial infarction, valvular heart disease or congestive heart failure.
    * Previous mediastinal radiotherapy.
    * Uncontrolled arterial hypertension despite optimal medical therapy.
    * Previous treatment with doxorubicin at cumulative doses in excess of 400 mg/m².
    * Symptomatic arrhythmia or any arrhythmia requiring treatment.
    * Abnormal ECG as detailed below:

      * QT interval prolongation:
      * QTc> 480 msec.
      * Left ventricular hypertrophy :
      * Sokolow Index: (R V5 or V6) + S V1)> 3.5mv.
      * Left bundle-branch block:
      * Complete: QRS> 0.12 sec. No Q wave is seen in leads V5 and V6. A notched R wave is seen in left leads and a notched S wave in right side leads.
      * Right bundle-branch block:
      * Complete: QRS> 0.12 sec. Secondary R (R') wave in leads V1-V2. Slurred S wave in leads D1 ,avL, V5 and V6.
      * Second-degree atrioventricular (av) block:
      * Mobitz I AV block, or Wenckebach block: Progressive prolongation of the PR interval causing progressive R-R interval shortening until a P wave fails to conduct the ventricle. The RR interval containing the blocked P wave is shorter than the sum of the twPP interval.
      * Mobitz II AV block is characterized by sudden unexpected blocked P waves without variation or prolongation of the PR interval. It can be 2:1, 3:1, 4:1 etc.
      * Third-degree atrioventricular block:
      * P waves and QRS complexes without mutual relationship. P wave rate is greater than that of QRS complexes.
      * Ischemia, injury and infarction:
      * Subendocardial ischemia. - Symmetrical T waves of increased amplitude.
      * Subepicardial ischemia. - Inverted symmetrical T waves.
      * Subendocardial injury. - ST segment depression (horizontal or descending).
      * Subepicardial injury. - ST segment elevation with upper convexity.
      * Infarction or necrosis. - Q wave voltage greater than 25% of R wave voltage.
      * Duration of Q wave is 0.04 sec or more
    * History of significant neurological or psychiatric disorders.
    * Active infection; infection by HIV, HBV or HCV. HIV, HBV or HCV testing are not required unless infection is clinically suspected.
    * Myopathy or any clinical situation that causes significant and persistent elevation of CK (> 2.5 ULN in two different determinations performed with one week apart).
    * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
    * Limitation of the patient's ability to comply with the treatment or follow-up protocol.
    * Uncontrolled endocrine diseases (e.g. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).
11. Known hypersensitivity to Aplidin®, mannitol, cremophor EL, or ethanol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celestia Higano, M.D., Principal Investigator — Seattle Cancer Care Alliance; Maha Hussain, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Aplidin®: Aplidin (Plitidepsin)
  Aplidin (plitidepsin): Aplidin® administered at a starting dose of 5 mg/m2, as a 3-hours intravenous infusion, every 2 weeks.
Period: Overall Study
Arm/Group | Aplidin®
Started | 8
Completed | 0
Not Completed | 8
Not completed — Progressive disease | 3
Not completed — Toxicity | 5

BASELINE CHARACTERISTICS:
Arm/Group | Aplidin®
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 60.5 [55.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With a ≥ 50% Prostate-specific Antigen (PSA) Decline Post-therapy
Time Frame: All patients were followed up to progressive disease, start of a new anti-cancer therapy, death or one year after the last treatment visit of the last patient, whichever occured first
Measure: Count of Participants; unit: Participants
Arm/Group | Aplidin®
Number analyzed (Participants) | 8
Participants
  PSA Progression | 1
  PSA Stabilization | 4
  PSA Progression NC | 2
  PSA Response NC | 1

2. Secondary Outcome: Objective Tumor Response According to RECIST
Description: Patients with an objective tumor response (complete response [CR] or partial response [PR]) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST), See Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, et al. New Guidelines to Evaluate the Response to Treatment in Solid Tumors. J Natl Cancer Inst 2000; 92:205-16.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aplidin®
Number analyzed (Participants) | 8
Participants
  stable disease | 4
  no response | 3
  non evaluable | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: To assess the antitumor activity of plitidepsin given intravenously over 3-hours every two weeks in patients with castrate metastatic adenocarcinoma of the prostate that have relapsed or progressed after 2 previous lines of systemic therapy, considering biological agents or chemotherapy as systemic therapy and taking into account that patients must have received prior docetaxel-based chemotherapy.
  PFS defined as time from the first day of study treatment to the day of a negative outcome (progression according to RECIST (Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, et al. New Guidelines to Evaluate the Response to Treatment in Solid Tumors. J Natl Cancer Inst 2000; 92:205-16) or death) or last contact. If any patient is lost to follow up before disease progression, the PFS will be censored at the date of the last tumor assessment. If there are no tumor assessments the patient will be censored at the first drug administration date.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aplidin®
Number analyzed (Participants) | 8
months | 1.76 [1.4 to 3.2]

4. Secondary Outcome: Overall Survival (OS)
Description: To assess the antitumor activity of plitidepsin given intravenously over 3-hours every two weeks in patients with castrate metastatic adenocarcinoma of the prostate that have relapsed or progressed after two previous lines of systemic therapy, considering biological agents or chemotherapy as systemic therapy and taking into account that patients must have received prior docetaxel-based chemotherapy.
  Survival is measured from the first day of study treatment to death or day of their last follow-up
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aplidin®
Number analyzed (Participants) | 8
months | 8.0 [5.7 to 9.8]

5. Secondary Outcome: Pain Improvement Rate
Description: To assess the antitumor activity of plitidepsin given intravenously over 3-hours every two weeks in patients with castrate metastatic adenocarcinoma of the prostate that have relapsed or progressed after two previous lines of systemic therapy, considering biological agents or chemotherapy as systemic therapy and taking into account that patients must have received prior docetaxel-based chemotherapy.
  Expressed as a change in pain intensity according to the pain intensity score on the 100 mm VAS (Visual Analogue Scale) and/or change in analgesic (morphine-equivalent mg) requirements after a pain stabilization period of 2-7 days
  Visual Analogue Scale (VAS), expressed in the pain intensity score on the 100 mm VAS scale (0=least possible pain to 100=worst possible pain)
Time Frame: 2-7 days for the pain stabilization required at baseline to ensure that baseline values are stable and reliable. The follow-up period was up to progressive disease, start of a new anti-cancer therapy, death or one year after the last treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Aplidin®
Number analyzed (Participants) | 8
units on a scale | 0 [-81.8 to 60.0]

6. Secondary Outcome: PSA Slope Between Baseline PSA Value and Nadir After the Start of Treatment
Description: To assess the antitumor activity of plitidepsin given intravenously over 3-hours every two weeks in patients with castrate metastatic adenocarcinoma of the prostate that have relapsed or progressed after two previous lines of systemic therapy, considering biological agents or chemotherapy as systemic therapy and taking into account that patients must have received prior docetaxel-based chemotherapy.
  It was calculated as (nadir value-baseline value)/(nadir date-baseline date). Modifications in the slope of PSA changes before and after the start of treatment with Aplidin will also be explored.
Time Frame: From baseline until progression or initiation of another anticancer therapy, death or one year after the last treatment visit of the last patient, whichever occurred first.
Population: One patient less because there were not PSA measurements after baseline
Measure: Median (Full Range); unit: ng/ml/days
Arm/Group | Aplidin®
Number analyzed (Participants) | 7
ng/ml/days | 1.3 [-1.9 to 23.8]

ADVERSE EVENTS:
Arm/Group | Aplidin®
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aplidin® (N=8)
Acute myocardial infarction (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Electrocardiogram ST-T change (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aplidin® (N=8)
Anaemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 8
Influenza like illness (General disorders) | 1
Injection site reaction (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Thirst (General disorders) | 1
Herpes zoster (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatine phosphokinase (Investigations) | 1
Blood creatinine (Investigations) | 2
Blood glucose (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 3
Haemoglobin (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Troponin increased (Investigations) | 1
Weight decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Claustrophobia (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Bladder pain (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Ischaemia (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days